CLINICAL TRIAL: NCT04700774
Title: Behavioral Activation for Depression: A Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Mia Skytte OToole, Associate professor, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BA Dep 20
Record Dates: First submitted 2020-12-21; First posted 2021-01-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to active treatment or a 10-week waitlist followed by active treatment (BA or mBA). The active treatment is also based upon randomization, where individuals will receive either standard BA or mBA, and will be followed for 6 months post treatment.
Who Masked: Participant
Masking Description: It will not be known to participants whether they receive standard BA or mBA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mBA (Experimental): Motor enhanced behavioral activation. 10 sessions.
  Interventions: Behavioral: Behavioral activation
- BA (Experimental): Standard behavioral activation. 10 sessions.
  Interventions: Behavioral: Behavioral activation
- Waitlist (No Intervention): 10 week waitlist.

INTERVENTIONS:
Behavioral: Behavioral activation — Brief Behavioral Activation Treatment with and without motor enhancement. All patients will receive 10 online video sessions. BA focuses on increasing overt behaviors to bring patients into contact with reinforcing environmental contingencies and corresponding improvements in thoughts, mood, and quality of life (Hopko, Lejuez, et al., 2003). BA follows the basic behavioral principles of extinction, shaping, fading, and in vivo exposure (Hopko & Lejuez, 2007; Lejuez et al., 2001, 2011). In the mBA condition only a) patients will be introduced to the idea that the motor system can be used in the service of action initiation and will receive an audio recording with motor manipulations to assist in action initiation and b) the therapist will conduct imaginary behavioral activation and - in session - complete questionnaires identical to those in the experiment before and after the bodily instructions presented in the treatment.
  Arms: BA; mBA

SUMMARY:
The present study is a randomized controlled trial that will evaluate two versions of behavioral activation (BA); one version which is a standard BA program and one which is a motor enhanced BA program (mBA). In both programs, the patient will receive all standard BA interventions, whereas these - in the mBA program - will be supplemented with interventions focused on noticing and manipulating posture and movement associated with action initiation. The mBA program builds upon recent evidence pointing to motor manipulations of posture and movement as having the potential to assist in action initiation and thus following through with the planned activity schedule. Previous research has shown that patient compliance with the activity schedule is causally associated with depression reduction, which will be explored as a mediator of treatment gains.

DETAILED DESCRIPTION:
Depression is a leading cause of disability worldwide (WHO, 2020). Nationally, more than 10.000 new cases of depression are registered each year with a higher frequency in women (Sundhedsstyrelsen, 2015). With depression comes reduced quality of life for the affected individual and a great economic burden for society. For instance, collectively, people with depression have more than 600.000 more visits to their general practitioner (GP) than people without depression, and when employed, they have 1.7 million more sick days than people without depression (Sundhedsstyrelsen, 2015). Access to effective treatment is thus crucial. Behavioral activation (BA) is an efficacious psychological treatment for depression; its effect may exceed that of medication and is equal to that of cognitive behavioral therapy (CBT) (Cuijpers, van Straten, & Warmerdam, 2007; Ekers et al., 2014). BA is therefore recommended as a first-line psychological treatment for mild to moderate depression by the National Institute for Health and Care Excellence (NICE CG90; 2009).

Depression is often described with reference to the disorder's cognitive characteristics, such as the depressogenic content of thoughts ( Beck, Rush, Shaw, & Emery, 1979) and the tendency to engage rumination and self-criticism (e.g., Mennin & Fresco, 2013) as well as behavioral characteristics such as lack of motivation, avoidance, and withdrawal (e.g., Lewinsohn, 1974). Although less commonly found in the description of depression, research has also documented bodily characteristics, including alterations to the motor system. Concerning the motor system, gait patterns associated with sadness and depression have been characterized by reduced walking speed, arm swing, and vertical head movements (Michalak et al., 2009). Successful treatment of depression thus may include - not only improvements in cognition and behavior - but also normalization of the motor system.

Although CBT and BA produce similar results in the treatment of depression, they are rooted in different theoretical models of depression. Traditional CBTs target the depressed individual's dysfunctional appraisals. They do so by inviting the client to restructure their thinking and expose themselves to situations that will help them in this endeavor. This is based on the assumption that the root of the problematic behavior in depression, first and foremost, is a result of dysfunctional thinking (e.g., "it doesn't matter anyway", "I will always be depressed") ( Beck et al., 1979). BA, on the other hand, is primarily rooted in a behavioral theory of depression. It builds on Lewinsohn's (1974) seminal work, holding that depression is the result of a loss or lack of response-contingent positive reinforcement, leaving the patient stuck in a maladaptive pattern of behavioral avoidance and withdrawal, preventing them from having rewarding interactions with their surroundings. In order to combat this avoidance and withdrawal behavior permeating depression, the patient in BA is invited to monitor their activities - mapping the dysfunctional patterns - and then to engage in activities that are important and joyful, if not at first, then over time (Lejuez, Hopko, Acierno, Daughters, & Pagoto, 2011; Martell, Dimidjian, & Herman-Dunn, 2010). Indeed, in the beginning, certain activities may not feel instantly rewarding, and the depressed person may only have a vague memory of a time when that activity was associated with joy. However, in BA, patients are invited to try to act 'outside-in', instead of 'inside-out', meaning that they refrain from acting according to their mood (low mood will likely lead to more avoidance and withdrawal behavior) and instead approach the planned activity regardless of their current mood (i.e., outside-in).

Previous research has shown that patient compliance with the activity schedule is causally associated with depression reduction (Ryba et al., 2014). Thus, theoretically and empirically, following through with the activity schedule presents as one of the most important mediators of treatment gains. However, patients may struggle with initiating the planned activities. In a sense, BA asks patients to do exactly the thing they feel like they cannot do, that is, get up and get going. Despite psychoeducation about the rationale of the treatment, and even when clients get initial experience with the fact that they feel better and more competent after a certain activity, they may still struggle with action initiation (Martell et al., 2010). Recent evidence points to motor manipulations of posture and movement as having the potential to be an important supplementary intervention within BA, enhancing the likelihood that clients follow through with the planned activity schedule. In a recent meta-analysis, we investigated the effect of motor manipulations (i.e., expansive/upright and contractive/slumped postures) on affective and behavioral outcomes. Across studies, we found that the manipulation of motor activity altered mood, emotions, and actions such that when individuals adopt neutral or expansive postures, they reported better mood, more positive emotions, and engaged in more approach behavior than when assuming contractive postures (Elkjær et al., 2020). These results could suggest that adopting neutral or expansive postures could be helpful for depressed individuals in initiating action.

Building on the solid findings from previous BA trials and the recent findings concerning the effects of motor manipulations, the present study is a randomized controlled trial that will evaluate two versions of BA, one version which is a standard BA program (Lejuez et al., 2011) and one which is a motor enhanced BA program (mBA). In both programs, the patient will receive all standard BA interventions, whereas these - in the mBA program - will be supplemented with interventions focused on noticing and manipulating posture and movement associated with action initiation. One hundred and seventeen individuals diagnosed with major depressive disorder (MDD) will be randomized to active treatment or a 10-week waitlist followed by active treatment. The active treatment is also based upon randomization, where individuals will receive either standard BA or mBA, and will be followed for 6 months post treatment. In the active treatment, individuals will receive 10 weekly video sessions, conducted using the secure and GDPR-approved video-conference program 'Zoom'.

Before and after the mBA program, patients will partake in an experiment. The effect of motor manipulations on responses to two different personally relevant emotional conflicts will be evaluated. One emotional conflicts will be one that is typical of those detected in depression, where an individual wishes they could or would enjoy approaching a situation but lack the motivation to do so (i.e., approach vs. withdrawal). The other will be one in which an individual wishes they could approach a situation but feel scared or nervous about doing so (approach vs. avoidance). Participants will be randomized to one of three experimental conditions: adopting expansive postures, contractive postures, or neutral postures. Effects will be evaluated concerning action tendencies, behavioral self-efficacy and experienced emotions. For the experiment taking place before treatment, patients will be compared to a group of matched healthy controls.

Hypotheses

It is hypothesized that 1) both BA and mBA will be more efficacious in reducing symptoms of depression than the waitlist, and 2) gains are expected to be maintained through the follow-up period.

It is also expected that 3) mBA with its extra treatment component focused on the motor system will be superior to BA of at least small magnitude (d=0.3; Bell et al., 2013). This added benefit of mBA is expected to be driven by compliance with the activity schedule as it is hypothesized 4) that the mBA condition can increase success with planned activities (i.e., quantity of completed activities and proportion of completed activities). 5) This success with planned activities is expected to mediate treatment gains in both BA and mBA.

Concerning the experiment, before treatment, 6) it is expected that depressed patients to show less approach behavior (i.e., less approach action tendencies, less behavioral self-efficacy, , and less positive emotions) in response to the emotional conflicts compared with healthy controls. Furthermore, 7) it is hypothesized that participants assuming neutral and expansive postures will respond with more approach behavior than participants adopting contractive postures. 8) Effects will be explored between groups (healthy vs clinical), thereby determining if the neutral and expansive motor displays are more or less facilitative of approach behavior, and if the contractive motor displays are more or less detrimental to such behavior, depending on clinical status. 9) Effects will also be explored comparing the two types of emotional conflicts.

Concerning the experiment following treatment, 10) it is expected that any differences between the healthy and clinical group detected at baseline will diminish or disappear, reflecting clinical improvement and normalization following treatment.

Collaborators:

Mai B. Mikkelsen, Gitte Tramm, Emme Elkjær, Kaj Sparle Christensen, Douglas S. Mennin, & Johannes Michalak

ELIGIBILITY:
Depressed participants:

Inclusion Criteria:

* A principal diagnosis of major depressive disorder (MDD) according to DSM-5 of a mild to moderate severity, that is, a 4 on a 0 (no depressive symptoms) to 8 (very severe symptoms) scale according to the ADIS-5 interview.
* Danish language proficiency.
* Ability and willingness to give informed consent.
* Be either non-medicated or stabilized [i.e., same dosage for a minimum of 8 weeks on antidepressant and antianxiety medication].
* Access to either a smartphone, tablet, or computer with video camera

Exclusion Criteria:

* Severe depression deemed to require more intense psychotherapy or medication.
* Non-stabilized medication (see above).
* A history of bipolar disorder.
* Current or past psychosis.
* Substance abuse or dependence judged to require treatment.
* Suicide risk requiring immediate hospitalization.
* Receiving any other current psychotherapy or counseling.

Healthy participants:

Will only be considered for participation if they can read and understand the Danish language and deemed able and willing to give informed consent. They will undergo diagnostic interviewing to ensure the absence of a current psychiatric diagnosis and the absence of a history of bipolar disorder or psyhosis according to the ADIS-5. They will also be excluded if they receive any psychotropic medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms (PHQ-9) | Change from pre to post (10 weeks) active treatment.
  Patient Health Questionnaire-9 (Spitzer et al., 1999; Spitzer et al., 2000)

SECONDARY OUTCOMES:
Depressive symptoms (PHQ-9) | Change from pre-treatment through 6-months follow-up
  Patient Health Questionnaire-9 (Spitzer et al., 1999; Spitzer et al., 2000)
Number of recovered patients in BA/mBA vs. waitlist | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  Number cacluated according to the minimal clinically important difference for the PHQ-9 (i.e., 5 score points; Lowe, Unutzer, Callahan, Perkins, & Kroenke, 2004)
Number of patients having obtained a reliable change in depressive symptoms in BA/mBA vs. waitlist | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  Calculated according to the reliable change index (Jacobsen & Truax, 1999) for the PHQ-9.
Exposure to environmental rewards (EROS) | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  The Environmental Reward Observation Scale (Armento & Hopko, 2007)
Intereoceptive awareness (MAIA) | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  The Multidimensional Assessment of Interoceptive Awareness, Version 2 (Mehling, Acree, Stewart, Silas, & Jones, 2018)
Behavioral activation and inhibition (BIS/BAS) | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  BIAS/BAS (Carver & White, 1994)
Perceived coping ability(CSES) | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  The Coping Self-Efficacy Scale (Chesney, Neilands, Chambers, Taylor, & Folkman, 2006
Rumination (RRS) | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  The Ruminative Response Scale, brooding subscale (Treynor, Gonzalez, & Nolen-Hoeksema, 2003)
Worry (PSWQ) | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  The Penn State Worry Questionnaire (Meyer, Miller, Metzger, & Borkovec, 1990)
Decentering (EQ) | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  The Experiences Questionnaire Decentering subscale (Fresco et al., 2007)
Dysfunctional attitudes (DAS) | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  Dysfuntional Attitude Scale SF1 (Beever et al., 2009; Weismann, 1979)
Quality of life (QoL) | Change form pre to post active treatment (10 weeks) and change from pre-treatment through 6-months follow-up
  The World Health Organization (WHO)-5 questionnaire

OTHER OUTCOMES:
PHQ-9 | Session by session change during the 10 weeks of active treatment
  Depressive symptoms will be evaluted session by session for mediation analyses
EROS | Session by session change during the 10 weeks of active treatment
  Environmental rewards will be evaluted session by session for mediation analyses
CSES | Session by session change during the 10 weeks of active treatment
  Coping ability will be evaluted session by session for mediation analyses
RRS | Session by session change during the 10 weeks of active treatment
  Ruminaiton will be evaluted session by session for mediation analyses
Activity log (kept by therapist) | Session by session change during the 10 weeks of active treatment
  Quantity and proportion of activities will be calculated for mediation analyses
EQ | Session by session change during the 10 weeks of active treatment
  Decentering ability will be tested as a competing mediator
DAS | Session by session change during the 10 weeks of active treatment
  Dysfunctional attitudes will be tested as a competing mediator
Overall activity level | Session by session change during the 10 weeks of active treatment
  Total steps taken (measured by pedometer) and exercise each day will be tested as a competing mediator
Perceived importance of activity | Change from pre to post experimental manipulation (10 minutes) (pre-treatment only for healthy participants, pre- and post-treatment for depressed participants)
  "How important is the activity to you?". Outcome in experiment (7-point Likert scale from 1 to 7)
Expected effect of activity on mood | Change from pre to post experimental manipulation (10 minutes) (pre-treatment only for healthy participants, pre- and post-treatment for depressed participants)
  "How do you expect the activity to affect your mood?" Outcome in experiment (7-point Likert scale from -3 [negative] to +3 [positive])
Perceived self-efficacy concerning activity | Change from pre to post experimental manipulation (10 minutes) (pre-treatment only for healthy participants, pre- and post-treatment for depressed participants)
  "How confident do you feel about your ability yo take the activity?". Outcome in experiment (7-point Likert scale from 1 to 7)
Perceived difficulty of completing activity | Change from pre to post experimental manipulation (10 minutes) (pre-treatment only for healthy participants, pre- and post-treatment for depressed participants)
  "How difficult is it for you to do the activity". Outcome in experiment (7-point Likert scale from 1 to 7)
Degree of avoidance and withdrawal motivation concerning activity | Change from pre to post experimental manipulation (10 minutes) (pre-treatment only for healthy participants, pre- and post-treatment for depressed participants)
  Withdrawal: "I do no feel like or have the energy to complete the activity." Avoidance: "I am scared, nervous or worried about doing the activity". Outcome in experiment (7-point Likert scale from 1 to 7)
Action tendencies (DAT; O'Toole & Mikkelsen, 2020) concerning activity | Change from pre to post experimental manipulation (10 minutes) (pre-treatment only for healthy participants, pre- and post-treatment for depressed participants)
  Outcome in experiment (8 drawings rated on a 5-point Likert scale from 1 to 5)
Negative and positive emotions when thinking about doing activity | Change from pre to post experimental manipulation (10 minutes) (pre-treatment only for healthy participants, pre- and post-treatment for depressed participants)
  8 negative and 7 positive emotions used as outcome in experiment (5-point Likert scale from 1 to 5)
State rumination (Brief State Rumination Inventory [BRSI]; Marchetti, Mor, Chiorri, & Koster, 2018) | Obtained post experiment only
  Outcome in experiment (statements rated from 0 to 100)

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University - Institute of Psychology and Behavioral Sciences, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/74/NCT04700774/SAP_000.pdf